CLINICAL TRIAL: NCT04940598
Title: Telehealth High Intensity Interval Exercise and Cardiometabolic Health in Spinal Cord Injury
Brief Title: High Intensity Interval Exercise SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Gordon Fisher, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 000526083; R21NR019309 (NIH)
Record Dates: First submitted 2021-06-16; First posted 2021-06-25 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Spinal Cord Injuries; Cardiometabolic Diseases
Keywords: High Intensity Interval Training; Telehealth Exercise; Armcrank Exercise; SCI
MeSH Terms: conditions — Spinal Cord Injuries | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: In a longitudinal study design, 40 participants with chronic SCI will be randomly assigned to one of the two study groups (HIIT and control) in a 1:1 ratio. Randomization will be performed using the block randomization method, Randomization will be performed using the block randomization method. A randomization list will be generated and assignments will be placed into closed envelopes and given to each study participant. Participants will be assessed at baseline and 16-wks post HIIT or control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval exercise (Experimental): High intensity interval arm crank exercise
  Interventions: Other: high intensity interval exercise
- No-Exercise Control (Other): No-exercise control group
  Interventions: Other: No-exercise control group

INTERVENTIONS:
Other: high intensity interval exercise — HIIT training will be delivered two times per week for 16 weeks (32 sessions). Each session will be separated by at least 24-hrs. Participants will be allowed to choose the days and times that they feel exercise will fit into their schedule. The HIIT protocol will be determined based on peak anaerobic power measures during an arm crank Wingate Cycle test. HIIT will consist of 20 minutes of exercise consisting of four minutes of arm crank exercise at 5% of peak anaerobic power followed by 30 seconds at 30% of the peak anaerobic power; this cycle will be repeated four times, ending with two minutes of recovery at 5% of peak anaerobic power.
  Arms: High intensity interval exercise
Other: No-exercise control group — No-exercise control group
  Arms: No-Exercise Control

SUMMARY:
This study will determine if the implementation of a home-based telehealth high intensity interval exercise-training (HIIT)program can significantly improve cardiometabolic health and physical function in a cohort of individuals with longstanding spinal cord injury (SCI). Results from this study will determine feasibility, overall enjoyment, and health impact of implementing a home-based telehealth HIIT program in individuals with SCI.

DETAILED DESCRIPTION:
For individuals with spinal cord injury (SCI), exercise participation reduces the risk of developing chronic cardiometabolic diseases, which are leading causes of rehospitalization and death within this population. Accordingly, recent SCI exercise guidelines have highlighted a need for exercise trials that can improve cardiometabolic factors such as glucose tolerance, blood lipids, blood pressure, and body composition. However, to date, the number of exercise trials examining these cardiometabolic outcomes in SCI is low, and these exercise regimens are often inconvenient for individuals with SCI to perform within their community. In addition to the functional impairment associated with the disability, individuals with SCI experience a number of barriers to exercise participation, such as lack of time (e.g. conflict with work schedule), accessible or usable equipment and facilities, and transportation. Thus, it is important to identify effective modes of exercise that can improve overall health but do not require a significant overall weekly time commitment. Investigators recently demonstrated that individuals with SCI could safely perform high intensity interval training (HIIT) using arm crank cycling and that as few as two days per week of HIIT could improve cardiometabolic health. Despite the advantages of HIIT, it is important to identify methods of implementing exercise trials that can successfully reach and maintain participation in larger cohorts. Recent work by the investigative group demonstrated that individuals with SCI expressed favorable perceptions of home-exercise training that incorporated telehealth technology, which allowed a fitness specialist to remotely monitor participants' training progress in real-time and provide verbal support via videoconferencing. This method of training holds even greater value for home-exercise programs that require monitoring to dose-specific protocols such as HIIT. However, the long-term success of HIIT will greatly depend on the ease at which the program can be implemented, as well as participants' adherence and perceptions of using the technology, which has not been investigated in SCI. The goal of this study is to integrate a home-based telehealth HIIT arm crank exercise training program in individuals with SCI and assess changes in cardiometabolic health and physical function. The secondary goal is to explore the uptake and implementation of HIIT in SCI. 40 participants will be randomized to home-based HIIT exercise or a no-exercise control group for 16-weeks. Body composition, aerobic fitness, muscular strength, and changes in cardiometabolic health will be assessed at baseline and 16-weeks post training. In addition to changes in cardiometabolic health outcomes, the investigators will also conduct interviews with participants to determine overall perceptions of the program, program likes and dislikes, perceived satisfaction and value, usability of equipment and technology, and factors that influence adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, 19-65 years of age.
2. Confirmed diagnosis of traumatic SCI at the cervical or thoracic level (C7-T12), classified as A, B, C, or D (motor and sensory complete or incomplete) on the AIS scale.
3. At least 6 months post-injury.
4. Able to independently operate an arm ergometer.
5. Have access to a wireless internet connection.
6. Medically stable, able to provide informed consent.

Exclusion Criteria:

1. Cardiovascular or renal diseases.
2. Pregnant women
3. Orthopedic conditions that prevents arm ergomtery
4. Upper extremity musculoskeletal conditions that prevents arm ergometry.
5. Neurological disorder that prevents arm ergometry
6. Participation in a structured exercise program currently or in the past 3 months.
7. Unable to perform exercise interventions

   -

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Fisher, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Adams J, Lai B, Rimmer J, Powell D, Yarar-Fisher C, Oster RA, Fisher G. Telehealth high-intensity interval exercise and cardiometabolic health in spinal cord injury. Trials. 2022 Aug 4;23(1):633. doi: 10.1186/s13063-022-06585-2. PMID 35927708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were identified by a computer-generated list of patients who are enrolled in the UAB SCI Model System and the Lakeshore Foundation Member Database and currently reside in the greater Birmingham, Alabama area. All potential participants were mailed a letter which describes the study, invites them to participate. Additional recruiting was done by posting fliers at the UAB Spain Rehabilitation Center (SRC) and Lakeshore Foundation.
Period: Overall Study
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Intensity Interval Exercise | No-Exercise Control | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (11.6) | 56.4 (8.1) | 52.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: inches] | 69.7 (2.9) | 66.7 (6.4) | 68.6 (4.4)
Body Weight [Mean (Standard Deviation); unit: kg] | 87.2 (23.7) | 94.3 (30.9) | 89.9 (24.7)
VO2 Peak [Mean (Standard Deviation); unit: ml/kg/min] | 11.6 (2.9) | 10.1 (.99) | 11 (2.4)
Insulin Sensitivity [Mean (Standard Deviation); unit: matsuda] | 3.5 (1.8) | 6.1 (4.2) | 4.5 (2.9)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 179.2 (36) | 178 (4.3) | 178.8 (27.4)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 132.6 (46.3) | 126.3 (30) | 130.2 (38.7)
HDL [Mean (Standard Deviation); unit: mg/dl] | 45.6 (6.9) | 51.7 (.58) | 47.9 (6.1)
LDL [Mean (Standard Deviation); unit: mg/dl] | 107 (30.4) | 101.1 (9) | 104.8 (23.6)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dl] | 95.2 (3.5) | 148.3 (85.6) | 115.1 (53.4)
Fasting Insulin [Mean (Standard Deviation); unit: mIU/L] | 10.6 (4.3) | 7.6 (4.1) | 9.5 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Aerobic Capacity Baseline
Description: All subjects will undergo a progressive peak oxygen assessment to determine aerobic capacity at the Lakeshore Foundation Exercise Physiology Facility. Subjects will be instructed to perform arm crank ergometer (Lode) at 10W for 2 min. Every 2 min thereafter, power output will be increased by 10W until voluntary fatigue. Peak aerobic power will be defined as VO2 at the point of failure to maintain 60-65 rotations per minute.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Number analyzed (Participants) | 5 | 3
ml/kg/min | 11.6 (2.9) | 10 (.99)

2. Primary Outcome: Aerobic Capacity Week 16
Description: as for outcome 1
Time Frame: 16weeks post training
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Number analyzed (Participants) | 5 | 3
ml/kg/min | 13.6 (2.2) | 9.9 (2.5)

3. Primary Outcome: Matsuda Index Baseline
Description: Oral glucose tolerance test. Following an overnight fast each subject will consume a 75g oral glucose load within 5 min. Blood samples will be collected immediately before and 60, 90, and 120 min following glucose ingestion for measurement of serum glucose and serum insulin. Insulin sensitivity was calculated using glucose and insulin values by the Matsuda Index, in which a higher number demonstrates an improvement in insulin sensitivity,
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Number analyzed (Participants) | 5 | 3
score on a scale | 3.5 (1.8) | 6.1 (4.2)

4. Primary Outcome: Matsuda Index Week 16
Description: as for outcome 3
Time Frame: 16weeks post training
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Number analyzed (Participants) | 5 | 3
score on a scale | 5.3 (3.5) | 6.5 (5.9)

5. Primary Outcome: Cholesterol Baseline
Description: Laboratory analyses. Concentrations of blood lipids will be determined in the Core Laboratory of the CCTS, NORC, and DRC.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Number analyzed (Participants) | 5 | 3
mg/dl | 179.2 (36) | 178 (4.4)

6. Primary Outcome: Cholesterol Week 16
Description: as for outcome 5
Time Frame: 16weeks post training
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Number analyzed (Participants) | 5 | 3
mg/dl | 193.8 (49.5) | 188 (25.3)

7. Primary Outcome: Body Composition Baseline
Description: Dual-energy X-ray absorptiometry (DXA). Percent Body Fat
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: Percent Fat
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Number analyzed (Participants) | 5 | 3
Percent Fat | 42.4 (1.1) | 47.5 (6.8)

8. Primary Outcome: Body Composition Week 16
Description: Dual-energy X-ray absorptiometry (DXA). Percent Body Fat
Time Frame: 16weeks post training
Measure: Mean (Standard Deviation); unit: Percent Fat
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Number analyzed (Participants) | 5 | 3
Percent Fat | 41.9 (2.8) | 46.9 (7.2)

9. Primary Outcome: Triglycerides Baseline
Description: as for outcome 5
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Number analyzed (Participants) | 5 | 3
mg/dl | 132.6 (46.3) | 126.3 (30.1)

10. Primary Outcome: Triglycerides Week 16
Description: as for outcome 5
Time Frame: 16-weeks post
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Number analyzed (Participants) | 5 | 3
mg/dl | 122.8 (39.1) | 102.3 (44.3)

11. Primary Outcome: HDL Baseline
Description: as for outcome 5
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Number analyzed (Participants) | 5 | 3
mg/dl | 45.6 (6.9) | 51.7 (0.6)

12. Primary Outcome: HDL Week 16
Description: as for outcome 5
Time Frame: 16-weeks post training
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Number analyzed (Participants) | 5 | 3
mg/dl | 52 (9.6) | 57.7 (8)

13. Primary Outcome: LDL Baseline
Description: as for outcome 5
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Number analyzed (Participants) | 5 | 3
mg/dl | 107.1 (30.4) | 101.1 (8)

14. Primary Outcome: LDL Week 16
Description: as for outcome 5
Time Frame: 16-weeks post training
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
Number analyzed (Participants) | 5 | 3
mg/dl | 117.5 (48.1) | 109.7 (22)

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | High Intensity Interval Exercise | No-Exercise Control
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/3

LIMITATIONS AND CAVEATS:
Limitations in this study include a small sample size. We were only able to recruit a total of 5 participants for this study, we had 5 participate in the exercise group and 3 in the control group. We modified the protocol at the end of year 2 to enable a wait-listed control group that would allow those assigned to the control condition the option to participate in the exercise arm of the study as well. COVID made it difficult to enroll participants for the first 2 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT04940598/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT04940598/ICF_001.pdf